CLINICAL TRIAL: NCT06680388
Title: Exploratory Clinical Study to Evaluate the Safety and Efficacy of Autologous CD19 CAR-T in the Treatment of Relapsed/Refractory Autoimmune Diseases
Brief Title: CD19 CAR-T in the Treatment of Relapsed/Refractory Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024072
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- patients with relapsed/refractory moderately or severely active systemic lupus erythematosus (SLE) (Experimental): Drug：CD19 CAR-T
  Interventions: Drug: Drug：CD19 CAR-T
- relapsed/refractory active diffuse cutaneous systemic sclerosis (dcSSc) (Experimental): Drug：CD19 CAR-T
  Interventions: Drug: Drug：CD19 CAR-T
- relapsed/refractory antineutrophil cytoplasmic antibody (ANCA) -associated vasculitis (AAV) (Experimental): Drug：CD19 CAR-T
  Interventions: Drug: Drug：CD19 CAR-T
- relapsed/refractory idiopathic inflammatory myopathy (IIM) (Experimental): Drug：CD19 CAR-T
  Interventions: Drug: Drug：CD19 CAR-T
- relapsed/refractory Sjogren 's syndrome (SS) (Experimental): Drug：CD19 CAR-T
  Interventions: Drug: Drug：CD19 CAR-T

INTERVENTIONS:
Drug: Drug：CD19 CAR-T — A total of 3 dose groups were set, with dose group 1 as the starting dose, which was performed according to the traditional 3 + 3 design rule as a single intravenous infusion.

SUMMARY:
Autoimmune diseases such as systemic lupus erythematosus (SLE), diffuse cutaneous systemic sclerosis (dcSSc), antineutrophil cytoplasmic antibody (ANCA) -associated vasculitis (AAV), idiopathic inflammatory myopathy (IIM), and Sjogren's syndrome (SS) have complex etiologies and are prone to cause systemic multiple organ damage. Because patients need lifelong medication due to repeated disease recurrence, and the current treatment of the above autoimmune diseases has limited efficacy and greater side effects, so that patients bear an excessive burden of disease, therefore, there is an urgent need to explore safer and more effective treatment.

Several autologous CAR-T products targeting CD19 have been marketed for the treatment of B-cell hematological malignancies. Depletion of B cells to suppress abnormal immune responses is also currently one of the popular strategies for the treatment of antibody-mediated autoimmune diseases, and many clinical studies of CAR-T against autoimmune diseases are still ongoing.

Therefore, a dose escalation trial is planned to evaluate the safety, tolerability, and preliminary efficacy of autologous CD19 CAR-T in patients with relapsed/refractory autoimmune diseases.

DETAILED DESCRIPTION:
This study is a single-center, open, exploratory clinical trial designed to evaluate the safety and efficacy of autologous CD19 CAR-T in the treatment of relapsed/refractory autoimmune disease.

The study will adopt the traditional dose escalation model "3+3" design, set up 3 dose groups, with 0.5×10^6 CAR+T cells /kg as the initial dose to increase, observe DLT, and conduct a 24-month safety and efficacy follow-up after cell infusion to observe the safety of autologous CD19 CAR-T. At the same time, preliminary efficacy evaluation was carried out.

ELIGIBILITY:
Inclusion Criteria:

* 1、aged 18 to 65 years (including 18 and 65 years), male or female;
* 2、Special criteria for different indications:
* 2.1 Subjects with relapsed/refractory moderate to severe SLE must meet the following criteria:
* 1) diagnosis of SLE according to the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria for SLE;
* 2) positive antinuclear antibody (ANA) (titer ≥ 1:80), and/or positive anti-dsDNA -antibody, and/or positive anti-Sm antibody at screening;
* 3) moderate to severe activity is defined as: SLEDAI-2000 ≥ 8 points at screening; if there is a score of low complement and/or anti-dsDNA antibody, the score for clinical symptoms of SLEDAI-2000 (except low complement and/or anti-ds-DNA antibody) needs to be ≥ 6 points;
* 4) stable standard treatment regimen for at least 6 months in the history of SLE before screening, and the disease remains active for at least 2 months before screening. Standard treatment regimen refers to stable use of any of the following drugs (alone or in combination): glucocorticoids (≤ 20 mg/day prednisone or equivalent), antimalarials (hydroxychloroquine ≤ 400 mg/day, chloroquine ≤ 500 mg/day), non-steroidal anti-inflammatory drugs (NSAIDs), biologics (rituximab, belimumab, tatacept) and other immunosuppressive agents or immunomodulators, including mycophenolate mofetil (≤ 2 g/day), azathioprine (≤ 2 mg/kg/day), methotrexate (≤ 20 mg/week);
* 2.2 Subjects with relapsed/refractory dcSSc were required to meet the following criteria:
* 1) diagnosis of SSc according to the 2013 EULAR/ACR classification criteria for systemic sclerosis (SSc);
* 2) diffuse cutaneous manifestations according to the 1988 LeRoy et al criteria, ie, extensive skin fibrosis with proximal elbow and/or knee skin involvement;
* 3) interstitial lung disease (ILD) at screening, and 45% predicted ≤ forced vital capacity (FVC) ≤ 70% predicted, or 40% predicted ≤ diffusing capacity for carbon monoxide (DLCO) ≤ 70% predicted;
* 4) relapse/refractory was defined as failure to respond to prior conventional therapy or relapse after disease remission. Conventional therapy was defined as the use of corticosteroids, cyclophosphamide, and at least 1 immunosuppressive/modifying agent for ≥ 6 months, including azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, rituximab, belimumab, and taitacept;
* 5) activity was defined as having at least 1 of the following: evidence of skin progression at screening, ie, an increase in mRSS score of ≥ 10% within the past 6 months; evidence of any of the following ILD activities at screening: newly diagnosed ILD within the past 6 months; decline in FVC of 10%, or decline in FVC of 5% with DLCO of 15% within the past 6 months in subjects with preexisting ILD.
* 2.3 Subjects with/refractory AAV must meet the following criteria:
* 1) a clinical diagnosis of granulomatous vasculitis (GPA) and microscopic polyangiitis (MPA) as defined by the 2012 Chapel Hill Consensus Conference (CHCC);
* 2) at least one major item or at least three other items in Birmingham Vasculitis Activity Score (BVAS) version 3;
* 3) positive antiproteinase-3 (PR3-ANCA) antibody or antimyeloperoxidase (MPO-ANCA) antibody at screening;
* 4) relapsed/refractory as defined by: Subjects with relapsed AAV: initial response to prior treatment with corticosteroids combined with immunosuppressive agents (cyclophosphamide, rituximab, azathioprine, methotrexate, mycophenolate mofetil, etc.) for at least 3 months (BVAS score 0 and glucocorticoid dose ≤ 7.5 mg/day prednisone or other equivalent glucocorticoid agents) or 1 - 2 additional items emerging in two consecutive assessments),Patients with relapsed disease within 12 weeks before screening; subjects with refractory AAV: those who had not achieved response after at least 3 months of previous treatment with glucocorticoids combined with immunosuppressive agents (cyclophosphamide, rituximab, azathioprine, methotrexate, mycophenolate mofetil, etc.) (BVAS score of 0 and glucocorticoid dose ≤ 7.5 mg/d prednisone or other equivalent glucocorticoid drugs);
* 2.4 Subjects with relapsed/refractory IIM were required to meet the following criteria:
* 1) have a ≥ 55% probability of being diagnosed with IIM according to the 2017 EULAR/ACR classification criteria for IIM, and were classified as having dermatomyositis (DM), polymyositis (PM), or immune-mediated necrotizing myopathy (IMNM) based on age at first onset, skin and muscle strength performance, laboratory tests, and muscle biopsy characteristics:；
* 2) disease activity/severity meeting the following criteria: free-hand muscle strength test-8 (MMT-8) score ≤ 141 (total score 150)；meet at least 2 of the other CSMs abnormalities: overall disease activity assessed by the patient [based on visual analogue scale (VAS)] score ≥ 2 points (range 0 - 10 points); overall disease activity VAS score ≥ 2 points (range 0 - 10 points) assessed by the physician; VAS score ≥ 2 points (range 0 - 10 points) for extramuscular overall disease activity assessed by the physician; Physician assessed health assessment questionnaire disability index (HAQ-DI) score ≥ 0.25 (range 0-3). At least 1 muscle enzyme level > 1.5 times the upper limit of normal (ULN).
* 2.5 Subjects with relapsed/refractory SS were required to meet the following criteria:
* 1) diagnosis of SS according to the 2016 EULAR/ACR classification criteria for SS;
* 2) anti-Ro/SSA antibody positivity at screening;
* 3) dynamic total salivary flow rate ≥ 0.05 mL/min or static total salivary flow rate ≥ 0.01 mL/min at screening;
* 4) activity was defined as: Sjögren 's Syndrome Disease Activity Index (ESSDAI) score ≥ 5 on 8 subitems;
* 3. The above autoimmune diseases that are intolerant to glucocorticoids and at least one other immunosuppressive agent or modulator or have insufficient efficacy in the past require: at least 3 months of treatment with glucocorticoids and at least two immunosuppressive agents (azathioprine, methotrexate, mycophenolate mofetil, etc.) at known effective doses;
* 4. good organ function:
* 1) blood routine: absolute neutrophil count (ANC) ≥ 0.5 × 109/L, platelet count (PLT) ≥ 20 × 10^9/L, hemoglobin ≥ 60 g/L;
* 2) coagulation function: international normalized ratio (INR) ≤ 1.5 times ULN, and activated partial prothrombin time (APTT) ≤ 1.5 times ULN;
* 3) liver function: serum aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3 times upper limit of normal (ULN), total bilirubin ≤ 1.5 times ULN;
* 4) renal function: serum creatinine ≤ 1.5 × ULN or creatinine clearance (Cockcroft Gault formula) ≥ 30 mL/min;
* 5) cardiac function: New York Heart Association (NYHA) grade I or II, and echocardiography (ECHO) left ventricular ejection fraction (LVEF) ≥ 50%, no pericardial effusion; 12-lead electrocardiogram (ECG) no clinically significant abnormal findings;
* 6) Pulmonary function: oxygen saturation ≥ 92% in non-oxygenated state under indoor ventilation; no clinically significant pleural effusion;
* 5. Expected survival greater than 6 months;
* 6. Subjects with partners of childbearing potential agree to use effective contraceptive measures throughout the treatment period and 24 months after treatment, while not donating eggs/sperm for assisted reproduction; female subjects of childbearing age (women who have undergone sterilization surgery or menopause ≥ 12 months are not considered to be of childbearing potential) have a negative urine pregnancy or blood pregnancy test during the screening period;
* 7. Voluntarily participate in this trial and sign the informed consent form. Exclusion Criteria
* 1. patients with previous or concurrent other active malignancies, including tumor-associated polymyositis/dermatomyositis. Cured or at least 2 years without recurrence of cervical carcinoma in situ, non-invasive basal cell or squamous cell skin cancer or radical treatment of local prostate cancer, ductal carcinoma in situ after radical resection;
* 2. combined with severe lung disease in the past 3 months, such as moderate to severe pulmonary hypertension (mean pulmonary arterial pressure > 60 mmHg by echocardiography), oxygen therapy with oxygen mask or non-invasive or invasive ventilator-assisted respiration during screening;
* 3. IgA, IgG, IgM below the lower limit of normal (LLN) at screening;
* 4. patients who have used any of the following drugs or treatments within the specified time:
* 1) B cell depletion therapy within 1 month before screening and no treatment failure as assessed by clinicians, including targeted CD20, CD22, CD52, CD38, BCMA monoclonal antibody or bispecific antibody;
* 2) high-dose human intravenous immunoglobulin within 1 month before screening; -3) Use of therapeutic doses of glucocorticoids (prednisone ≥ 20 mg/day or equivalent doses of other corticosteroids) within 24 hours before Qinglin pretreatment;
* 4) Has received corticosteroid pulse therapy (defined as doses ≥ 500 mg/day prednisone or equivalent doses of other corticosteroids) within 2 weeks;
* 5) has received taitacept within 2 weeks prior to Screening or belimumab within 3 weeks;
* 5. Patients with a history of severe central nervous system disease or related symptoms (excluding trigeminal nerve disease alone) in the past 6 months, including but not limited to: lupus encephalopathy, cerebrovascular disease, encephalitis, brain injury, aneurysm, cerebellar disease, organic brain syndrome, Parkinson's disease and other central nervous system diseases, as well as epilepsy, convulsions, aphasia, dementia and other symptoms;
* 6. Lupus crisis occurred within 3 months before screening, such as active central nervous system lupus, severe hemolytic anemia, severe thrombocytopenic purpura, severe granulocytopenia, severe myocardial injury, severe lupus pneumonia or pulmonary hemorrhage, severe lupus hepatitis, severe vasculitis, etc.;
* 7. Patients with severe kidney disease: severe lupus nephritis within 8 weeks before screening [defined as urine protein > 4g/24 hours or serum creatinine > 1.5 × ULN or creatinine clearance (Cockcroft Gault formula) < 30 mL/min;], or active nephritis requiring the use of drugs prohibited by the regimen, or requiring prednisone greater than 500 mg/d or other effective treatment for ≥ 14 days;
* 8. Patients who are severely allergic to the Qinglin pretreatment drugs used in this study and any component of autologous CD19 CAR-T;
* 9. hepatitis B surface antigen (HBsAg) positive and peripheral blood HBV DNA positive; hepatitis C virus (HCV) antibody positive and HCV RNA positive; treponema pallidum antibody positive; HIV antibody positive;
* 10. the presence of uncontrolled fungi, bacteria, viruses or other infections that are not suitable for participation in the study as assessed by the investigator;
* 11. history of major organ transplantation (such as heart and lung);
* 12. active tuberculosis or latent tuberculosis (defined as tuberculin skin test or interferon test positive, and no clinical symptoms or imaging evidence) at screening; -13. any of the following cardiovascular diseases (including but not limited to) occurred within 6 months before screening:
* 1) congestive heart failure, myocardial infarction, unstable angina pectoris, coronary angioplasty, stenting, coronary artery/peripheral artery bypass grafting;
* 2) severe arrhythmia requiring treatment (such as persistent ventricular tachycardia, ventricular fibrillation, torsades de pointes, etc.); congenital long QT syndrome, left anterior hemiblock (bifascicular block), asymptomatic right bundle branch block into the study;
* 3) Uncontrolled hypertension (systolic blood pressure greater than 160 mmHg and/or diastolic blood pressure greater than 100 mmHg), history of hypertensive crisis or hypertensive brain;
* 14. combined with other autoimmune diseases (including but not limited to eosinophilic granulomatous polyangiitis, cryoglobulinemia vasculitis, inclusion body myositis, anti-glomerular basement membrane disease, Behcet 's disease or Takayasu' s arteritis, etc.) in addition to the target indications requiring systemic treatment;
* 15. with a family history of non-IIM such as drug-induced myopathy, human immunodeficiency virus-related myopathy;
* 16. pregnant or lactating women;
* 17. vaccinated with live vaccine within 6 weeks before clear lymphocyte pretreatment;
* 18. participated in other interventional clinical studies within 3 months before signing the informed consent form, received active investigational drug treatment, or intentionally participated in another clinical trial or received autoimmune diseases other than those specified in the protocol throughout the study;
* 19. patients with depression or suicidal mental illness;
* 20. researchers believe that there are other factors that are not suitable for inclusion or affect the subject 's participation or completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT); | within 28 (+3) days after receiving the infusion.
  • Grade ≥ III acute GvHD that has not resolved to Grade I or II within 7 days, with the exception of acute GvHD with skin involvement only; • Grade ≥ 4 CRS, or Grade 3 CRS that has not resolved to Grade 1 or 2 within 14 days of onset; • Grade 4 ICANS or Grade 3 ICANS lasting ≥ 7 days; • Other Grade 3 or higher AEs associated with autologous CD19 CAR-T and lasting ≥ 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: wang ying, Principal Investigator — wangying1@ihcams.ac.cn
Locations (1):
- Chinese Academy of Medical Sciences Hospital of Hematology (Chinese Academy of Medical Sciences Institute of Hematology), Tianjin, 300020, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No